CLINICAL TRIAL: NCT00990327
Title: The ASPECT Trial: A Phase III, Randomized, Double-Blind Crossover Trial of Apadenoson for the Detection of Myocardial Perfusion Defects Using Single-Photon Emission Computed Tomography (SPECT) Myocardial Perfusion Imaging (MPI)
Brief Title: Study of the Safety and Efficacy of Apadenoson for Detection of Myocardial Perfusion Defects Using SPECT MPI
Acronym: ASPECT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PGX-III-AP-001
Record Dates: First submitted 2009-10-02; First posted 2009-10-06 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Myocardial Perfusion Imaging
MeSH Terms: conditions — Coronary Artery Disease | interventions — ATL 146e; Adenosine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Apadenoson (Experimental): In period 1, subjects will receive a clinically-indicated rest/stress gated SPECT-MPI with adenosine. In period 2, subjects will receive a rest/stress gated SPECT-MPI with apadenoson or the active comparator: adenosine.
  Interventions: Drug: Apadenoson SPECT-MPI; Drug: Adenosine SPECT-MPI
- Adenosine (Active Comparator): In period 1, subjects will receive a clinically-indicated rest/stress gated SPECT-MPI with adenosine. In period 2, subjects will receive a rest/stress gated SPECT-MPI with apadenoson or the active comparator: adenosine.
  Interventions: Drug: Apadenoson SPECT-MPI; Drug: Adenosine SPECT-MPI

INTERVENTIONS:
Drug: Apadenoson SPECT-MPI — Apadenoson single bolus IV injection 100 or 150 ug
  Other Names: DPC-A78445-00, DPH-068645-01, ATL146e, DWH 146e
Drug: Adenosine SPECT-MPI — Single IV infusion for 6 minutes at a rate of 140 µg/kg body weight per minute.
  Other Names: Adenoscan

SUMMARY:
The purpose of this study is to see whether apadenoson is as effective as adenosine when used as a pharmacological stress agent in myocardial SPECT-Imaging to detect defects in the supply of blood to the heart muscle (myocardial perfusion defects). The study will also look at whether apadenoson is better tolerated than adenosine when used in SPECT-MPI.

DETAILED DESCRIPTION:
Adenosine is an effective vasodilator used in SPECT-Myocardial Perfusion Imaging (SPECT-MPI). However, it produces transient symptoms that are poorly tolerated by most subjects. PGxHealth has designed a multi-center, randomized crossover, double-blind study to compare the safety and effectiveness of apadenoson to adenosine (Adenoscan®) in SPECT-MPI. Subjects who are clinical candidates for SPECT-MPI will be enrolled to undergo two sequential SPECT-MPI studies. The first study will use adenosine as the stress agent in approximately 1300 subjects. Eligible subjects will then be randomized in a 1:2 assignment ratio to receive a second SPECT-MPI using either adenosine or apadenoson as the pharmacologic stress agent, with the goal of obtaining a total of 753 subjects who complete both studies. The similarity of the results from the two adenosine:adenosine stress tests will be compared to those from the adenosine:apadenoson tests to assess efficacy. The incidence and intensity of commonly reported side effects will be compared to evaluate improved tolerability.

ELIGIBILITY:
Inclusion Criteria:

* High pretest probability of CAD based on the ACC/AHA guidelines for relative risk, or past medical h/o CAD

Exclusion Criteria:

* Ingestion of a caffeinated or methylxanthine food substance (e.g. chocolate, cocoa) within 24 hours before receiving apadenoson or adenosine
* Treatment with dipyridamole within 24 hours, or theophylline, aminophylline, or pentoxifylline within 72 hours (or 4 half-lives, whichever is longer) prior to receiving apadenoson or adenosine
* Acute MI, new onset of ischemia or PCI within 30 days prior to SPECT-MPI at either Period 1 or Period 2; or CABG within 90 days prior to SPECT-MPI at either Period 1 or Period 2
* Active severe asthma or severe chronic obstructive pulmonary disease (COPD) which, in the Investigator's opinion, places the subject at risk for severe bronchoconstriction
* History or evidence of clinically significant cardiac condition and rhythm disorder, in the absence of a functioning permanently implanted pacemaker
* Hemodynamically significant valvular disease, outflow tract obstruction, or uncontrolled severe hypertension
* Current significant medical, surgical, psychiatric, or other illness or pathology that could potentiate any adverse pharmacological event associated with an investigational drug
* Subject with past medical history of hepatitis B or C, or recent hepatitis A
* Pretreatment hypotension (systolic BP < 90 mm Hg) or tachycardia (HR > 100 bpm)
* Known history of cerebral vascular accident or suspected transient ischemic attack within 30 days prior to signed informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 863 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Presence of myocardial perfusion defect as based on SPECT-MPI | Up to 2 hours after study drug administration in Period 1 and 2

SECONDARY OUTCOMES:
Incidence and patient rated intensity of most commonly reported side effects (e.g. dyspnea, flushing, chest pain, headache) associated with use of adenosine compared to apadenoson in SPECT-MPI | 1 hour after Period 2 study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: David B Bharucha, MD, PhD, FACC, Study Director — Forest Laboratories
Locations (122):
- United States (103):
  - Forest Investigative Site 152, Birmingham, Alabama
  - Forest Investigative Site 250, Mobile, Alabama
  - Forest Investigative Site 223, Phoenix, Arizona
  - Forest Investigative Site 191, Phoenix, Arizona
  - Forest Investigative Site 230, Jonesboro, Arkansas
  - Forest Investigative Site 153, Little Rock, Arkansas
  - Forest Investigative Site 108, La Mesa, California
  - Forest Investigative Site 111, Mission Viejo, California
  - Forest Investigative Site 234, Murrieta, California
  - Forest Investigative Site 146, Roseville, California
  - Forest Investigative Site 225, Sacramento, California
  - Forest Investigative Site 122, Sacramento, California
  - Forest Investigative Site 105, Santa Rosa, California
  - Forest Investigative Site 196, Walnut Creek, California
  - Forest Investigative Site 132, Hartford, Connecticut
  - Forest Investigative Site 102, Newark, Delaware
  - Forest Investigative Site 205, Daytona Beach, Florida
  - Forest Investigative Site 233, Edgewater, Florida
  - Forest Investigative Site 164, Gainesville, Florida
  - Forest Investigative Site 120, Jacksonville, Florida
  - Forest Investigative Site 198, Jacksonville, Florida
  - Forest Investigative Site 118, Jacksonville, Florida
  - Forest Investigative Site 124, Jacksonville, Florida
  - Forest Investigative Site 125, Jacksonville, Florida
  - Forest Investigative Site 126, Jacksonville Beach, Florida
  - Forest Investigative Site 180, Melbourne, Florida
  - Forest Investigative Site 183, Miami, Florida
  - Forest Investigative Site 106, Miami, Florida
  - Forest Investigative Site 201, Naples, Florida
  - Forest Investigative Site 240, Tampa, Florida
  - Forest Investigative Site 238, Wellington, Florida
  - Forest Investigative Site 155, Augusta, Georgia
  - Forest Investigative Site 199, Cumming, Georgia
  - Forest Investigative Site 204, Tucker, Georgia
  - Forest Investigative Site 116, Honolulu, Hawaii
  - Forest Investigative Site 137, Boise, Idaho
  - Forest Investigative Site 138, Boise, Idaho
  - Forest Investigative Site 227, Chicago, Illinois
  - Forest Investigative Site 228, Joliet, Illinois
  - Forest Investigative Site 173, Winfield, Illinois
  - Forest Investigative Site 113, Indianapolis, Indiana
  - Forest Investigative Site 168, Valparaiso, Indiana
  - Forest Investigative Site 171, West Des Moines, Iowa
  - Forest Investigative Site 133, Overland Park, Kansas
  - Forest Investigative Site 248, Crestview Hills, Kentucky
  - Forest Investigative Site 241, Owensboro, Kentucky
  - Forest Investigative Site 202, Alexandria, Louisiana
  - Forest Investigative Site 257, Covington, Louisiana
  - Forest Investigative Site 114, Auburn, Maine
  - Forest Investigative Site 107, Scarborough, Maine
  - Forest Investigative Site 109, South Portland, Maine
  - Forest Investigative Site 193, Baltimore, Maryland
  - Forest investigative Site 197, Westminster, Maryland
  - Forest Investigative Site 143, Detroit, Michigan
  - Forest Investigative Site 207, Petoskey, Michigan
  - Forest Investigative Site 177, Saint Louis Park, Minnesota
  - Forest Investigative Site 131, Tupelo, Mississippi
  - Forest Investigative Site 176, Kansas City, Missouri
  - Forest Investigative Site 159, St Louis, Missouri
  - Forest Investigative Site 188, Missoula, Montana
  - Forest Investigative Site 115, Albany, New York
  - Forest Investigative Site 212, Buffalo, New York
  - Forest Investigative Site 165, Kingston, New York
  - Forest Investigative Site 224, Manhasset, New York
  - Forest Investigative Site 139, Massapequa, New York
  - Forest Investigative Site 208, Raleigh, North Carolina
  - Forest Investigative Site 249, Sanford, North Carolina
  - Forest Investigative Site 214, Fargo, North Dakota
  - Forest Investigative Site 235, Akron, Ohio
  - Forest Investigative Site163, Columbus, Ohio
  - Forest Investigative Site 161, Columbus, Ohio
  - Forest Investigative Site 156, Lorain, Ohio
  - Forest Investigative Site 185, Sandusky, Ohio
  - Forest Investigative Site 101, Westlake, Ohio
  - Forest Investigative Site 182, Oklahoma City, Oklahoma
  - Forest Investigative Site 190, Bend, Oregon
  - Forest Investigative Site 217, Portland, Oregon
  - Forest Investigative Site 213, Camp Hill, Pennsylvania
  - Forest Investigative Site 154, Philadelphia, Pennsylvania
  - Forest Investigative Site 134, Philadelphia, Pennsylvania
  - Forest Investigative Site 218, Philadelphia, Pennsylvania
  - Forest Investigative Site 160, Pittsburgh, Pennsylvania
  - Forest Investigative Site 187, Sellersville, Pennsylvania
  - Forest Investigative Site 117, Wyomissing, Pennsylvania
  - Forest Investigative Site 149, Charleston, South Carolina
  - Forest Investigative Site 172, Simpsonville, South Carolina
  - Forest Investigative Site 229, Spartanburg, South Carolina
  - Forest Investigative Site 167, Johnson City, Tennessee
  - Forest Investigative Site 192, Johnson City, Tennessee
  - Forest Investigative Site 128, Amarillo, Texas
  - Forest Investigative Site 252, Grapevine, Texas
  - Forest Investigative Site 200, McKinney, Texas
  - Forest Investigative Site 181, Plano, Texas
  - Forest Investigative Site 253, San Antonio, Texas
  - Forest Investigative Site 186, Sugar Land, Texas
  - Forest Investigative Site 231, Tomball, Texas
  - Forest Investigative Site 232, Tomball, Texas
  - Forest Investigative Site 236, Provo, Utah
  - Forest Investigative Site 210, Charlottesville, Virginia
  - Forest Investigative Site 110, Roanoke, Virginia
  - Forest Investigative Site 151, Seattle, Washington
  - Forest Investigative Site 142, Spokane, Washington
  - Forest Investigative Site 144, Madison, Wisconsin
- Brazil (19):
  - Forest Investigative Site 306, Salvador, Estado de Bahia
  - Forest Investigative Site 307, Curitiba, Paraná
  - Forest Investigative Site 308, Belo Horizonte - MG
  - Forest Investigative Site 317, Brasília - DF
  - Forest Investigative Site 311, Campinas
  - Forest Investigative Site 313, Curitiba
  - Forest Investigative Site 305, Curitiba
  - Forest Investigative Site 314, Curitiba - PR
  - Forest Investigative Site 316, Niterói
  - Forest Investigative Site 309, Passo Fundo - RS
  - Forest Investigative Site 318, Porto Alegre - RS
  - Forest Investigative Site 310, Porto Alegre - RS
  - Forest Investigative Site 315, Rio de Janeiro
  - Forest Investigative Site 319, Rio de Janeiro - RJ
  - Forest Investigative Site 304, Rio de Janeiro - RJ
  - Forest Investigative Site 301, Salvador - BA
  - Forest Investigative Site 303, São José
  - Forest Investigative Site 302, São Paulo - SP
  - Forest Investigative Site 312, São Paulo - SP